CLINICAL TRIAL: NCT03644134
Title: A Personalized Intervention to Manage Physiological Stress and Improve Sleep Patterns in Obese Type 2 Diabetes Emirati Patients: a Randomized Controlled Clinical Trial.
Brief Title: A Personalized Intervention to Manage Physiological Stress and Improve Sleep Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Bashair Mussa, Assistant Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RashidCDR; University of Sharjah (Other: University of Sharjah)
Record Dates: First submitted 2018-08-18; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes, Physiological Stress, Sleep Pattern
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Assessment of physiological stress and sleep pattern intervention consists of (i) information session (ii) pre-assessment (first assessment) of stress and recovery levels, and sleep patterns (iii) individual feedback sessions and action plans based on the outcomes of the initial assessment (iv) monitoring and follow-ups (v) post-assessment (second assessment) of stress and recovery levels and sleep patterns
  Interventions: Behavioral: Assessment of physiological stress and sleep pattern
- Control Group (No Intervention): The control protocol only includes (i) information session (ii) pre-assessment (initial assessment and (iii) post-assessment (second assessment) of stress and recovery levels and sleep patterns.

INTERVENTIONS:
Behavioral: Assessment of physiological stress and sleep pattern — The personalized intervention consists of (i) information session (ii) pre-assessment (first assessment) of stress and recovery levels, and sleep patterns (iii) individual feedback sessions and action plans based on the outcomes of the initial assessment (iv) monitoring and follow-ups (v) post-assessment (second assessment) of stress and recovery levels and sleep patterns.
  Arms: Intervention Group

SUMMARY:
Globally, type 2 diabetes mellitus (DM) and obesity are considered to be the fastest growing disorders and their prevalence has increased dramatically over the last twenty years.

Recent studies have shown that about 19% of UAE population has been diagnosed with DM and 57% of Emirati patients with type 2 DM are obese.

Optimal glycemic control and weight management involve comprehensive lifestyle approaches including nutrition recommendations and adequate levels of physical activity.

However, recent views have suggested that there are other factors, such as sleep deprivation and stress, contribute to development of type 2 DM.

Taking into account the previous findings, the present study was designed to investigate the effects of a personalized intervention on weight and glycemic control in Emirati patients with type 2 DM. The intervention involves assessment and modification of sleep patterns and stress levels.

DETAILED DESCRIPTION:
The present study is a randomized controlled trial which was conducted at Rashid Centre for Diabetes and Research (RCDR) in Ajman which in one of the seven Emirates of the United Arab Emirates (UAE). The study was approved by the research ethics committee of Al Qassimi Clinical Research Centre, Al Qassimi Hospital (Ministry of Health, UAE).

The study population is comprised of Emirati individuals (n = 51) who attending RCDR diabetes clinics in a quarterly basis (an initial visit and three follow-up visits per annum). The participants were recruited from RCDR diabetes clinics and through different methods including (i) direct contact (ii) distribution of informative flyers and (iii) phone calls using Diamond, an electronic medical database of RCDR patients. The screening process involved 110 Emirati patients with T2DM and 51 individuals were eligible to participate in the present trial based on the following inclusion and exclusion criteria. The inclusion criteria were (i) Age between 18-60 years (ii) Body Mass Index (BMI > 25 Kg/m2) and (iii) T2DM. The exclusion criteria were (i) Age < 18 and > 60 years (ii) BMI < 25 Kg/m2) (iii) type 1 DM (iv) diagnosis of atrial fibrillation and/or atrial flutter and/or bundle branch block and (v) heart transplantation.

The eligible participants were randomly allocated into an intervention group (n = 26) and or into a control group (n = 25). Non-compliance was the main obstacle to maintain the same number of the randomized participants in each group and 19% and 24 % of the participants in the intervention and control group, respectively, did not attend the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years
* Body Mass Index (BMI > 25 Kg/m2)
* T2DM

Exclusion Criteria:

* Age < 18 and > 60 years
* BMI < 25 Kg/m2)
* Type 1 DM
* Diagnosis of atrial fibrillation and/or atrial flutter and/or bundle branch block heart transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2015-07-14 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 6 months
  Measurement of body weight at the site visit pre/post the intervention
Change in BMI | 6 months
  Measurement of BMI at the site visit pre/post the intervention
Change in HbA1c | 6 month
  Measurement of HbA1c at the site visit pre/post the intervention

IPD SHARING:
Plan to Share IPD: No